CLINICAL TRIAL: NCT01252576
Title: Linguistic and Cultural Validation in Italian of Female Sexual Function Index Questionnaire (FSFI)
Brief Title: Linguistic and Cultural Validation in Italian of Female Sexual Function Index (FSFI) Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Club Italiano Femminile di Urologia (Other)
Collaborators: Società Italiana di Urologia (SIU) (Other)
Responsible Party: D.ssa Donata Villari, CIFU
Other Study IDs: 1-Villari
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Sexual Dysfunction
Keywords: FSFI; female sexual function; italian validation
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- women with and without sexual dysfunction: women with and without female sexual dysfunction

SUMMARY:
300 italian women will be enroll for linguistic and cultural validation in italian of Female sexual function index (FSFI). This questionnaire is used in most countries to investigate female sexual function. To date there are not validate questionnaires in italian on female sexual function. We decided to start the validation process to give a validated tool to italian investigators.

DETAILED DESCRIPTION:
A linguistic translation from the original language into the target language (Italian) will be carried out in parallel by two independent, native Italian-speaking professional translators, with English as their first foreign language. A first consensus meeting, which will involve the two translators and the research group, to compare the Italian versions and yielded a first-consensus Italian version of the scale. After this first phase the study will conduct in multiple Italian centres located in Northern, Central and Southern Italy. At each centre, the FSFI will administer to a female population of subjects with and without sexual dysfunction. Women will be administer the questionnaire at baseline and 2 weeks later, so as to evaluate the test-retest reliability. The patients will ask whether encountered any difficulty (ease of completion, comprehension, problems, etc). The number of patients who will encounter problems in correctly understanding questions and precoded answers will be recorded and discussed. Will also ask the women to indicate the way to ameliorate the test, and, if possible, the changes will be performed. A back-translation of the Italian consensus version will be carried out by a native American English-speaking professional translator, with Italian as her first foreign language, to control the adherence of translation with the original one. The final Italian version of the FSFI will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-65 years

Exclusion Criteria:

* mental diseases that do not permit to understand questionnaire

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women from general population whit or without sexual dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Test-retest reliability of FSFI italian translation | 15 days
  Test-retest reliability of professional translation in italian language of female sexual function index test.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Teresa Filocamo, MD, Principal Investigator — Club Italiano Femminile di Urologia
Locations (1):
- SS Annunziata Hospital, Savigliano, Cuneo, Italy